CLINICAL TRIAL: NCT00297180
Title: A Double-Blind, Randomized, Placebo-controlled Study to Evaluate Weight Loss, Safety, Tolerability and Pharmacokinetics in Obese Subjects Following 12-Week Dosing of GW869682, an SGLT2 Inhibitor
Brief Title: Weight Loss In Obese Subjects Taking Either GW869682 Or Placebo 3 Times Per Day For 12 Weeks
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: KGO105858
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Obesity
Keywords: hunger; obesity; sodium-dependent glucose transporter; GW869682; body composition; SGLT2 inhibitor; weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW869682

SUMMARY:
GW869682 causes glucose to be excreted in the urine. The purpose of this study is to see whether enough calories from glucose are excreted in the urine to cause weight loss.

ELIGIBILITY:
Inclusion criteria:

* Have a BMI within range 30.0 to 40.0kg/m2, inclusive.
* Females who meet above criteria must be physiologically incapable of becoming pregnant (ie., surgically sterilized, or post-menopausal per protocol definition).

Exclusion criteria:

* History of eating disorders.
* Recent history of weight loss or gain.
* Had gastrointestinal surgery for treatment of obesity.
* Type 1 or type 2 diabetes mellitus.
* Have a positive urine drug screen.
* Have liver disease.
* Have hepatitis B, hepatitis C, or HIV antibodies.
* Have a thyroid disorder that is not under control with medication.
* Have any disease (such as heart, liver, blood, nervous system, or kidney disease, or cancer).
* Are unable to participate in an exercise program.
* Have used weight loss drugs within 3 months before the start of the study.
* Are currently using warfarin, digoxin, oral anti-coagulants (other than aspirin and non-steroidal anti-inflammatory drugs), oral or injectable corticosteroids (inhaled & intranasal corticosteroids are permitted), or antiretroviral medications.
* Used of any investigational drug or device during the study or within 30 days prior to 1st dosing of study medication.
* High or low blood pressure.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2006-01; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Percentage change in body weight from baseline to Week 12. | from baseline to Week 12.

SECONDARY OUTCOMES:
Blood levels of GW869682 at the Week 2 and Week 11. | at the Week 2 and Week 11

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Portland, Oregon